CLINICAL TRIAL: NCT03230968
Title: Reduction in Morbidity, Complications and Mortality Caused by Respiratory Diseases Using a Personalized Integral Model of Care.
Brief Title: Use of a Respiratory Care Model in Population Older Than 15 Years in Orizaba, Veracruz Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Edith Elizabeth Ferreira Guerrero, Epidemiologist, Instituto Nacional de Salud Publica, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CI:1026; SALUD-2010-01-140645 (Other Grant/Funding Number: CONACYT)
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Disease
Keywords: Practical Approach to Lung Health; Respiratory diseases; Mexico
MeSH Terms: conditions — Respiration Disorders; Respiratory Tract Diseases | interventions — Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 without intervention (No Intervention): In selected heath centers we interviewed all consenting patients older than 15 years. Before the physician consultation, we investigated sociodemographic, epidemiologic, clinical characteristics and reason for seeking health services. Immediately after consultation, we asked the patient his/her diagnoses. We confirmed all diagnoses with treating physicians. If the patient had been diagnosed with respiratory disease, we collected information on prescribed treatment, and classified the type of respiratory disease and comorbidities based on the 10th International Classification of Diseases (ICD-10). Patients were given follow up one month later.
- Phase 2 with intervention (Active Comparator): We trained health personnel from the participating health centers on implementation of the proposed model based on the AIRE guidelines previously approved by the AIRE committee of the National Institute for Respiratory Diseases. The AIRE guidelines have been adapted from WHO "Practical Approach to Lung Health". Once the model was in action we interviewed all consenting patients older than 15 years as in phase 1.
  Interventions: Behavioral: Integral Action Program for Respiration

INTERVENTIONS:
Behavioral: Integral Action Program for Respiration
  Arms: Phase 2 with intervention

SUMMARY:
Background. Mexico is lacking guidelines that provide an integral approach for the prevention and control of respiratory diseases in adults. The World Health Organization (WHO) proposed a "Practical Approach to Lung Health" (PAL) using generic guidelines to be used in primary health care settings for diagnosis and treatment of respiratory diseases. These guidelines were adapted to the Mexican context as AIRE campaign by the Instituto Nacional de Enfermedades Respiratorias, Mexico. Objective. To evaluate the feasibility and effectiveness of implementing a model of care for respiratory diseases in adults based on AIRE guidelines,. Materials and methods. Prospective quasi-experimental pre-post study. During 03-08/2013 (phase 1), investigators recruited consenting subjects older than 15 years of age seeking medical care in primary care centers in Orizaba, Veracruz. Researchers investigated sociodemographic, epidemiological and clinical information before consultation. On patients who had been diagnosed with respiratory disease by a physician, researchers investigated prescribed treatment on leaving the physician´s office. A month later conducted a home visit to investigate clinical outcome. During 09/2014 we trained doctors from the participating health centers in "AIRE" guidelines. From 10/2014 to 03/2015 (phase 2) researchers again surveyed all consenting subjects older than 15 years of age who received health services in the same health centers following the same procedures as in phase 1.

DETAILED DESCRIPTION:
The design was that of a prospective quasi-experimental pre-post study. A pre-survey and a follow-up survey were used.Investigators selected 4 health centers in the Sanitary Jurisdiction in Orizaba, Veracruz, two located in rural areas (Potrerillo and Tlilapan) and two located in urban areas (Río Blanco and Orizaba). The pre-survey (phase1) was conducted on all consenting individuals older than 15 years seeking health services in selected health centers. Before the physician consultation, researchers investigated sociodemographic, epidemiologic, clinical characteristics and reason for seeking health services. Immediately after consultation, researchers asked the patient his/her diagnoses. Investigators confirmed all diagnoses with treating physicians. If the patient had been diagnosed with respiratory disease, researchers collected information on prescribed treatment, and classified the type of respiratory disease and comorbidities based on the 10th International Classification of Diseases (ICD-10). Researchers conducted a home visit one month after the consultation to determine clinical evolution, occurrence of referral to a specialist, if the patient had obtained prescribed drugs at the health center or at a private drugstore and if the patients had been hospitalized.

During September 2014 researchers trained health personnel from the participating health centers on implementation of the proposed model based on the AIRE guidelines previously approved by the AIRE committee of the INER. The AIRE guidelines have been adapted from WHO "Practical Approach to Lung Health" and include management of asthma, acute respiratory infections (ARI, that comprises acute bronchitis and pneumonia), chronic obstructive pulmonary disease (COPD), infections of the upper respiratory airways, and preventive measures for smoking, tuberculosis and breathing disorders during sleep.

The model was presented to the authorities of the participating health services and of the local hospital (Regional Hospital in Río Blanco (HRRB, its acronym in Spanish) as well as to health personnel involved in treatment of respiratory diseases, to promote their participation, counseling and support for the referral and counter-referral of patients.

The implementation of the guidelines included: 1) availability of the guidelines for the management of respiratory diseases in primary care "AIRE", that were revised and modified based on the analysis of the first phase of the study. Physicians providing primary care in the health centers and at the local hospital revised the guidelines to ensure that language was understandable. 2) Distribution of educational materials to health personnel including printed and electronic versions of AIRE guidelines, algorithm for management of acute and severe respiratory disease, and operational and good clinical practices manuals; 3) Training at the INER of the pulmonologist of the local hospital on AIRE guidelines and certification in spirometry. 4) Development of two workshops for 97 physicians and nurses of the participating health centers on AIRE Guidelines, oximetry tests, spirometry, referral and counter-referral of patients and clinical cases with the participation of specialized physicians from the INER, HRRB and the Instituto Nacional de Salud Pública (INSP); 5) Creation of a respiratory health network between primary care facilities, hospital and public health offices.

Researchers considered that patients participated in one of the two phases according to the period in which they sought health services.

Researchers defined a patient with a respiratory disease as any patient who after consultation with a physician was diagnosed with a respiratory disease according to the ICD-10. The medical diagnosis was obtained from the patient and confirmed with the treating physician and classified according to ICD-10. Respiratory diseases were classified in the following categories: emphysema, asthma and bronchitis, allergic rhinitis, lung cancer, chronic bronchitis, COPD and TB. Researchers also used a second categorization as follows: viral infections, bacterial infections and chronic diseases following the national clinical practice guidelines . Comorbidities were classified in the following categories: diabetes, hypertension, HIV and heart disease. The reason for seeking medical attention was classified into 20 categories. Researchers defined timeliness in requesting of health services measuring the interval from the onset of symptoms to request of physician consultation both as a continuous variable and as a dichotomic variable using as cut off >3 days. Researchers obtained the physician prescription and classified prescribed drugs as antibiotics, corticosteroids, cough suppressants, expectorants, bronchodilators, analgesics and antihistamines. Researchers also grouped cough suppressants, expectorants, analgesics and antihistamines in one category.

Researchers categorized age in 3 groups: 15 to 44 years, 45 to 59 years and >60 years. The variable "type of floor" was classified in two categories (hard floor/earth floor) according to the material of the floor.

Smoking was categorized as whether the patient was a current smoker or not. Alcohol consumption was dichotomized in more or equal or less than 14 alcoholic drinks per week. Use of drugs was categorized as to whether the patient reported using drugs during the study period. Researchers considered a patient was exposed to dust or smoke if he/she had worked for more than a year in a place with dust, smoke or vapors. Researchers considered occupational exposure to asbestos if the patient had worked for more than a year in a place with asbestos. Biomass exposure was categorized as whether the patient was currently exposed or not.

Researchers compared sociodemographic, epidemiologic and clinical characteristics of patients demanding physician consultation and of patients who were diagnosed with respiratory disease according to study period. In the bivariate analysis researchers used U of Mann Whitney test for continuous variables that didn't follow a normal distribution, chi-squared of Pearson test for dichotomous variables and binomial test for categorical variables.

Researchers compared by bivariate analyses the following outcomes according to study phase: 1) Acquisition of prescribed drugs in the pharmacy of the health center; 2) Treatment based on guidelines; 3) Clinical outcome; 4) Referral to a specialist. Using multivariate unconditional logistic regression, we built three models to investigate the association between phase of the study and 1) Acquisition of prescribed drugs in the pharmacy of the health center; 2) Treatment based on guidelines; 3) Clinical outcome. Variables with p < 0.20 in the bivariate analysis and biological plausibility were included in multivariate models. Multivariate models were built considering patients as clusters given that each patient could have had more than one drug prescription. Researchers estimated the odds ratio (OR) and 95 per cent confidence intervals (95% CI), and identified the covariates that were independently associated with each outcome.

All statistical analyses were performed using the statistical package STATA V13.3 (StataCorp LP).

ELIGIBILITY:
Inclusion Criteria:

* People older than 15 years of age that go to one of the health clinics seeking medical attention for any cause.

Residency in the study site.

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of prescribed drugs acquired in the pharmacy of the health center as stated in the questionnaire | One month after physician consultation
  The variable was categorized in: health center (all the prescribed medication was obtained from the pharmacy in the health center), and other pharmacy and/or health center (all or a part of prescribed medication was obtained in private establishments)
Accordance of prescribed treatment (based on questionnaire) with proposed guidelines | One month after physician consultation
  For each respiratory disease patient we evaluated if he/she had received treatment in compliance to AIRE guidelines
Clinical outcome of each participant based on follow up questionnaire | One month after physician consultation
  Clinical outcome was classified as follows: cure (disappearance of signs and symptoms and patient described as "healthy"), improvement (improvement of signs and symptoms), drop out (the patient stopped taking prescribed medications despite continuing signs and symptoms), still on treatment or death.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ferreira, MD, Principal Investigator — Instituto Nacional de Salud Pública

IPD SHARING:
Plan to Share IPD: No